CLINICAL TRIAL: NCT01737541
Title: Fluoxetine for Motor Recovery After Acute Intracerebral Hemorrhage (FMRICH): a Randomised Placebo-controlled Trial
Brief Title: Fluoxetine for Motor Recovery After Acute Intracerebral Hemorrhage
Acronym: FMRICH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study recruitment was suspended due to lack of funding
Sponsor: Universidad Autónoma de Aguascalientes (Other)
Responsible Party: Principal Investigator, Juan Manuel Marquez-Romero, Profesor Investigador, Universidad Autónoma de Aguascalientes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 83/11
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Intracerebral Hemorrhage; Motor Impairment
Keywords: Cerebrovascular Disorders; Cardiovascular Diseases; Intracerebral Hemorrhage; Serotonin Uptake Inhibitors; Therapeutic Uses
MeSH Terms: conditions — Cerebral Hemorrhage; Cerebrovascular Disorders; Cardiovascular Diseases | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine (Experimental): fluoxetine per os 20 mg daily
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): per os daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine
  Other Names: Fluoxac
  Arms: Fluoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter clinical trial that will be carried out in Mexico. The purpose of this study is to test whether a 3-month treatment with fluoxetine enhances motor recovery in non-depressed patients with acute intracerebral hemorrhage.

DETAILED DESCRIPTION:
Spontaneous, nontraumatic intracerebral hemorrhage (ICH) is a subtype of stroke that causes a great amount of disability, economic and social burden. This is particularly true in developing countries where it accounts for between 20% and 50% of all strokes. Pharmacological and surgical interventions have been attempted to diminish the mortality and disability derived from ICH, with unsuccessful results. Recently the use of Fluoxetine in addition to physical rehabilitation has been proven useful to improve motor recovery from cerebral infarct. The purpose of this study is to test whether a 3-month treatment with fluoxetine enhances motor recovery in non-depressed patients with acute intracerebral hemorrhage.

This is a randomized, double-blind, placebo-controlled, multicenter clinical trial. This trial will recruit 86 patients with intracerebral hemorrhage of both sexes, ages >18 years, from four Mexican hospitals. The patients will receive either 20mg of fluoxetine or a placebo once daily for 90 days. The primary outcome is the mean change in Fugl-Meyer Motor Scale score between inclusion (day 0) and day 90. The secondary outcomes will be changes in Barthel Index, Modified Rankin scale and National Institutes of Health (NIH) Stroke Scale. The outcomes will be measured at day 45±7days and at day 90, for a total of four visits with each subject (at screening and at 0, 45 and 90days).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had an acute intracerebral hemorrhage within the past 10 days causing hemiparesis or hemiplegia
* Fugl-Meyer motor scale (FMMS) scores of 55 or less
* Written informed consent for participation in the trial

Exclusion Criteria:

* Severe post-stroke disability (National Institutes of Health stroke scale [NIHSS] score >20)
* Premorbid disability, evidenced by residual motor deficit from a previous stroke
* Comprehension deficit or severe aphasia
* Previous diagnosis of depression or one of the following:

  * Hospital Anxiety and Depression Scale score ≥11 points
  * Taking antidepressant drugs two weeks before inclusion
* Taking neuroleptic drugs or benzodiazepines two weeks before inclusion
* Other major diseases with life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Motor Scale score | Baseline and 90 days
  Change from Baseline in Fugl Meyer Motor Scale score at 90 days

SECONDARY OUTCOMES:
Barthel Index | Baseline and 90 days
  Change from Baseline in Barthel Index at 90 days
modified Rankin Scale | Baseline and 90 days
  Change from Baseline in modified Rankin Scale at 90 days
NIH Stroke Scale | Baseline and 90 days
  Change from Baseline in NIH Stroke Scale at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Marquez-Romero, MD, Principal Investigator — Universidad Autónoma de Aguascalientes; Angel A Arauz, PhD, Study Director — Instituto Nacional de Neurología y Neurocirugía
Locations (4):
- Mexico (4):
  - Hospital General de Zona #1, Aguascalientes, Aguascalientes
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Instituto Nacional de Neurología y Neurocirugía, Mexico City, Mexico City
  - Hospital Regional de Alta Especialidad Dr. Juan Graham Casasus, Villahermosa, Tabasco

REFERENCES:
- [Background] Marquez-Romero JM, Arauz A, Ruiz-Sandoval JL, Cruz-Estrada Ede L, Huerta-Franco MR, Aguayo-Leytte G, Ruiz-Franco A, Silos H. Fluoxetine for motor recovery after acute intracerebral hemorrhage (FMRICH): study protocol for a randomized, double-blind, placebo-controlled, multicenter trial. Trials. 2013 Mar 19;14:77. doi: 10.1186/1745-6215-14-77. PMID 23510124
- [Derived] Marquez-Romero JM, Reyes-Martinez M, Huerta-Franco MR, Ruiz-Franco A, Silos H, Arauz A. Fluoxetine for motor recovery after acute intracerebral hemorrhage, the FMRICH trial. Clin Neurol Neurosurg. 2020 Mar;190:105656. doi: 10.1016/j.clineuro.2019.105656. Epub 2019 Dec 28. PMID 31896491
- See also: Full text protocol — http://www.trialsjournal.com/content/14/1/77